CLINICAL TRIAL: NCT00954369
Title: A Phase 0, Open Label, Non-randomized, Multi-center, Exploratory and Safety Study of [F-18]W372
Brief Title: Exploratory and Safety Study of [F-18]W372
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: W372000
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; AD; W372; W372000; [F-18]W372; exploratory; imaging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F-18]W372 (Experimental): Approximately twenty (20) adult subjects including ten (10) healthy volunteers and ten (10) high probability AD subjects, as defined by protocol criteria
  Interventions: Drug: [F-18]W372

INTERVENTIONS:
Drug: [F-18]W372 — The individual doses of [F-18]W372 contain a maximum of 20 mCi for normal volunteers and 10 mCi for high probability AD subjects.
  The single IP dose is administered to the study subject immediately prior to the start of PET imaging.
  Other Names: [F-18] W372; W372

SUMMARY:
PHASE: Phase 0, Exploratory Study

OBJECTIVES: To collect drug safety, bio-distribution and dosimetry data, to begin collection of PET/CT imaging data, to acquire experience to improve study design and the conduct of future studies.

DESIGN: Exploratory, open label, non-randomized, multi-center study.

DURATION: Three visits - one screening, one imaging, and one follow-up visit at 24 hours post-dose

PROCEDURES: Informed consent, collection of demographic information and medical history, administration of mental status exam, physical examination, vital signs, 12-lead ECGs, routine blood tests to assess major organ functions, complete blood counts and clinical chemistries for safety, dosing with [F-18]W372, PET imaging scans of brain (in sixteen subjects), whole body PET imaging and urine collections for dosimetry evaluation (in four subjects only), observation and interviews following imaging to collect adverse events.

SUBJECTS: Twenty (20) subjects ≥ 55 years old:

Group 1 will consist of 10 subjects who have a low probability of being currently positive for Alzheimer's Disease (AD) as defined by the protocol criteria (MMSE ≥ 28). Four of the 10 subjects will undergo whole body PET imaging for dosimetry evaluations, and 6 of the 10 subjects will undergo PET imaging of the brain only.

Group 2 will consist of 10 subjects who have a high probability of currently being positive for AD as defined by the protocol criteria (MMSE < 24); these 10 subjects will undergo PET imaging of the brain only.

DETAILED DESCRIPTION:
[F-18]W372 is being developed as a diagnostic radiopharmaceutical for PET imaging of the human brain.

SMI is seeking to determine if [F-18]W372 might be useful as a noninvasive assessment tool in aid of clinical evaluations of subjects with conditions associated with increased amyloid-β deposits, such as Alzheimer's disease.

Compared to the other non-invasive imaging approach, the values of amyloid PET imaging are more sensitive and accurate than previously established measures by FDG PET or volumetric MRI for diagnostic classification of subjects, suggesting that amyloid PET ligands may be more useful in differentiating among Alzheimer's disease, mild cognitive impairment, and normal aging as well as other neurodegenerative diseases. Therefore, this novel kind of molecular markers may provide advantages to measure amyloid plaques in vivo, have the potential to revolutionize early diagnosis of Alzheimer's disease, and hopefully will facilitate the AD diagnosis with improved accuracy.

In this exploratory study, the novel PET ligand for imaging amyloid plaques will be evaluated in age-matched normals with low probability being AD and subjects with high probability being AD in order to determine the bio-distribution, visualize signal/background in brains, and ultimately evaluate the safety and feasibility of [F-18] W372 as a potential PET biomarker for imaging amyloids in human brains.

The IP presents no known risks from either in vitro study in cell lines or in vivo study in animals according to preclinical investigations of this compound.

The population to be studied consists of a total of approximately twenty adult subjects, which will be a two group assignment. Group one will consist of ten subjects who have a low probability of being currently positive for Alzheimer's disease (AD) as defined by the protocol criteria. Four of the ten subjects in Group one will undergo evaluations for dosimetry. Group two will consist of ten subjects who have a high probability of currently being positive for AD as defined by the protocol criteria.

In the first year, this exploratory trial will be conducted as a Phase 0 study designed to evaluate bio-distribution data, to collect baseline imaging data, and to gather preliminary safety data for this investigational product. Based on the analyzed study results, this information will be considered in the design of future clinical trials.

The primary objectives of this exploratory study are:

* To collect drug safety information, bio-distribution data, and radiation dosimetry estimation
* To evaluate the drug uptake and signal/background information in brain PET imaging for subjects having a high probability of being currently positive for AD and age-matched subject having a low probability of being currently positive for AD
* To use this exploratory Investigational New Drug (eIND) document in order to obtain the necessary information to file an IND (Investigational New Drug) application with the FDA (Food and Drug Administration)

The secondary objective for this exploratory study is:

• To begin collection of baseline PET imaging data and to gain information to improve the study design for the conduct of future trials

The trial is expected to begin subject enrollment in approximately August 2009 and end subject participation in approximately December 2009, depending on the rate of enrollment.

The subject is expected to attend several visits, adding up to several hours (about 10 hours) of participation over three visits: a screening visit (Visit 1 - about 2 hours), a PET/CT imaging visit (Visit 2 - about 3-4 hours), and a follow up visit (Visit 3 - about 1 hour) about 24 hours after receiving the investigational product.

The investigational product will be administered to each qualified subject via a bolus injection (approximately 10 mCi will be administered for all subjects, except 20 mCi for the four subjects with a low probability of being positive for AD that are involved in the dosimetry analysis). This dose will not exceed 20 mCi, as the imaging time will extend out to approximately three hours. A larger dose (20 mCi) is needed in order to obtain quality images at the later time points.

Each study subject study subject will undergo three (3) visits. Visit 1 will be an initial screening visit to obtain informed consent and to determine if the prospective subject meets inclusion / exclusion criteria by having eligibility blood labs drawn and assessing mental status by performing the Mini-Mental Status Exam (MMSE). Concomitant medications and adverse events are recorded from the time of informed consent through Visit 3. Visit 2 will be an imaging visit in which a physical exam is performed, vital signs are measured, ECG testing is done, and pre-dose blood labs are drawn for safety. The subject then receives one dose of investigational product and undergoes PET imaging. The subject will undergo additional vital sign measurements and ECG testing after dosing during Visit 2. Visit 3 will be done to repeat the drawing of blood labs for safety, measure vital signs, ECG testing is done. All three visits must be completed in order to complete participation in the study.

ELIGIBILITY:
Inclusion Criteria:

Low Probability Subjects for AD:

* Subject has reached his or her 55th birthday at the time of the investigational product administration, and is male or female of any race / ethnicity
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of communicating with study personnel
* For inclusion into Group 1, in the opinion of the Investigator, the subject has a low probability of being currently positive for AD that is determined by a Mini Mental State Examination (MMSE ≥ 28)

High Probability Subjects for AD:

* Subject has reached his or her 55th birthday at the time of the investigational product administration, and is male or female of any race / ethnicity
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of communicating with study personnel
* For inclusion into Group 2, in the opinion of the Investigator, the subject has a high probability of being currently positive for AD that is determined by a Mini Mental State Examination (MMSE < 24)

Exclusion Criteria:

For All Subjects:

* Subject is not capable of complying with study procedures
* Female subject is pregnant

  * Exclude non-post menopausal females as defined by being one year without menses, or cannot be pregnant from her past medical history
* Subject has prior history of stroke or other condition of the head or neck that, in the Investigator's opinion, might affect circulation to the head or image interpretation
* Subject has a medical condition associated with elevated amyloid levels, such as amyloid angiopathy, familial amyloidosis, chronic kidney dialysis, Down's syndrome
* Subject has a history of significant cerebrovascular disease
* Subject has a significant hepatic or renal disease as defined by previous medical history or abnormal hepatic and renal functions determined by lab results not within the following ranges, or, in the opinion of the Investigator, the values are not acceptable for the subject to be included:

  * Total bilirubin within 2x institutional upper limits of normal
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limits of normal
  * Serum creatinine ≤ 2x institutional upper limits of normal
  * BUN within 2x institutional upper limits of normal
* Subject has previously received [F-18]W372 at any time
* Subject has been involved in an investigative, radioactive research procedure within the past 14 days
* Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete data or data quality
* Subject has a history in the last five years of significant prescription or nonprescription drug or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety will be the outcome demonstrated in this clinical trial through analyses of adverse events in subjects who receive study drug. | Three (3) study visits, including the initial screening visit, the imaging visit, and the 24 hour follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Min-Ying Su, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States